CLINICAL TRIAL: NCT05586308
Title: Pilot Study of Incentive-based and Media Literacy-informed Approaches to Improve Vaping Cessation Among Young Adults
Brief Title: Incentive-based and Media Literacy Informed Approaches to Improve Vaping Cessation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0596-22-EP; U54GM115458 (NIH)
Record Dates: First submitted 2022-10-14; First posted 2022-10-19 (Actual); Results first posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-01

CONDITIONS: Behavior, Health Risk; Implementation Science; E Cigarette Use; Cessation, Smoking; Incentives; Engagement, Patient; Peer Support; Media Literacy
MeSH Terms: conditions — Health Risk Behaviors; Vaping; Smoking Cessation; Patient Participation

STUDY DESIGN:
Intervention Model Description: This study employs a pilot, 4-arm randomized clinical trial design.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Active control (Other): Participants in this arm will receive an evidence-based text-messaging support.
  Interventions: Behavioral: Text-massaging suport
- Media literacy (Active Comparator): Participants will receive media literacy e-learning lessons and an evidence-based text-messaging support.
  Interventions: Behavioral: Text-massaging suport; Behavioral: Media literacy
- Financial incentive (Active Comparator): Participants will receive financial incentive intervention and an evidence-based text-messaging support.
  Interventions: Behavioral: Text-massaging suport; Behavioral: Financial incentive
- Combined (Experimental): Participants will receive media literacy e-learning lessons, financial incentive, and an evidence-based text-messaging support program.
  Interventions: Behavioral: Text-massaging suport; Behavioral: Financial incentive; Behavioral: Media literacy

INTERVENTIONS:
Behavioral: Text-massaging suport — Text-messaging quitting support program (i.e., This is Quitting) is an evidence-based, free mobile program from Truth Initiative designed to help young people quit vaping. The program is fully automated and interactive. To establish or reinforce perceived social norms and social support around quitting, a majority of messages come from other users who have submitted them to the program.
Behavioral: Financial incentive — 1. Participants will earn $3 for each saliva cotinine sample submission regardless of positive or negative results after the quit day (an assessments at Week 6, Week 8, Week 10, and Week 12, during the abstinence phase)
  2. Participants will earn additional escalating rewards for each negative sample- $7 for Week 6, $12 for Week 8, $17 for Week 10, and $22 for Week 12 (2 months after the target quit date). The bonus starts at $7 and increase by $5 for each subsequent negative cotinine sample (i.e., $7, $12, $17, and $22).
  3. A reset contingency will be used. That is the reward amount will be returned back to original $7 if there is a missing or positive saliva cotinine sample
  Arms: Combined; Financial incentive
Behavioral: Media literacy — Media literacy e-learning lessons cover topics regarding what e-cigarettes are and how they work, how nicotine and nicotine addiction affects the brain and behavior, how to prepare to quit vaping, developing a quit plan and how to deal with cravings and relapse. The program focuses on changing knowledge, attitudes and beliefs related to e-cigarette use, as well as emphasizing vaping related media literacy.
  Arms: Combined; Media literacy

SUMMARY:
This study aims to evaluate the feasibility and compare the preliminary effect of vaping cessation program consisting of media literacy education and real-time text messaging support and leverage insights from behavioral economics to enhance social and financial incentives to improve program engagement, and eventually abstinence. Our hypotheses are that 1) the Combined arm is associated with improved vaping abstinence to the Media literacy and Financial incentive arms; and 2) the financial incentive-related arms (either Combined or Financial incentive) enhance engagement compared to the non-incentive related arms.

DETAILED DESCRIPTION:
The objective of this pilot study is to evaluate the feasibility and compare the potential effect of different vaping cessation intervention components in addition to evidence-based text-messaging support, including 1) media literacy interactive e-learning lessons, 2) financial incentives, and 3) combined (media literacy + financial incentive) on vaping abstinence among current young adult vapers over a three-month timeframe with the following specific aims: Aim 1. To assess the feasibility of a multi-component vaping cessation program; and Aim 2 To evaluate the preliminary effect of a multicomponent vaping cessation program. Eligible participants are young adults aged 19-29 and are current vapers (i.e., has vaped in the previous 30 days).We will employ a 4-arm, feasibility randomized trial design to determine the preliminary effect of different vaping intervention components on vaping abstinence over a 3-month timeframe, consisting of a 1-month quitting preparation phase and 2-month abstinence phase. Eligible participants (n=80) will be randomized (in a 1:1:1:1 ratio), using a computer-generated algorithm, to to one of four vaping cessation interventions: 1) Active control: text-messaging support, 2) Media literacy: media literacy + text-messaging support, 3) Financial incentive: financial incentive + text-messaging support, and 4) Combined: media literacy e-learning lessons + financial incentive + text-messaging support, at the baseline visit. Regardless of intervention arms, all enrolled participants will receive receive an evidence-base text-messaging support program for quitting vaping (This is Quitting). Participants will be followed through a 3-month study period including a 1-month quitting preparation phase and a 2-month abstinence phase. All participants will be asked to provide the 5 saliva cotinine samples- at baseline and end-of-study visits and 3 at video calls (remote submissions). Participants who assigned to the financial incentive Combined groups will be provided monetary rewards for submitting saliva cotinine samples during the abstinence period. To examine the feasibility of biomarker testing for toxic exposures, for a subsample of 20 participants, a panel of biomarkers of toxic exposures will be measured at baseline and at the end of study.

ELIGIBILITY:
Inclusion Criteria:

* Aged 19-29
* Report vaping in the previous 30 days
* Have access to internet/video chat/SMS text message
* Are interested in quitting vaping in the next 30 days

Exclusion Criteria:

* Must meet all the inclusion criteria
* Self-report as currently pregnant or planning to become pregnant in the next 3 months
* Already involved in vaping cession programs (either behavioral or medical intervention)

Ages: 19 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-12-07 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2025-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tzeyu Michaud, PhD, Principal Investigator — University of Nebraska
Locations (1):
- Unversity of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in vaping cessation program targeting youth/young adults. Data shared will be coded, with no PHI included. Approval of the request and execution of all applicable agreements (i.e. a data transfer/use agreement) are prerequisites to the sharing of data with the requesting party.
Supporting Information: SAP, ICF, CSR
Time Frame: Data requests can be submitted starting 12 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing/USE Agreement.

REFERENCES:
- [Derived] Michaud T, Puga T, Archer R, Theye E, Zagurski C, Estabrooks P, Dai HD. Enhancing Text Message Support With Media Literacy and Financial Incentives for Vaping Cessation in Young Adults: Protocol for a Pilot Randomized Controlled Trial. JMIR Res Protoc. 2025 Feb 21;14:e60527. doi: 10.2196/60527. PMID 39983103

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We worked with READi Core at the University of Nebraska Medical Center to first generate a list of potentially eligible participants, filtering for age and using smart text data to determine the vaping or smoking status. A study invitation email was sent to individuals on this potential participant list . In this email, interested individuals will be directed to complete web-based screening questions via REDCap to assess their eligibility.
Groups:
- Financial Incentive: Participants will receive financial incentive intervention and an evidence-based text-messaging support.
  Text-massaging suport: Text-messaging quitting support program (i.e., This is Quitting) is an evidence-based, free mobile program from Truth Initiative designed to help young people quit vaping. The program is fully automated and interactive. To establish or reinforce perceived social norms and social support around quitting, a majority of messages come from other users who have submitted them to the program.
  Financial incentive: 1. Participants will earn $3 for each saliva cotinine sample submission regardless of positive or negative results after the quit day (an assessments at Week 6, Week 8, Week 10, and Week 12, during the abstinence phase) 2. Participants will earn additional escalating rewards for each negative sample- $7 for Week 6, $12 for Week 8, $17 for Week 10, and $22 for Week 12 (2 months after the target quit date). The bonus starts at $7 and increase by $5 for each subsequent negative cotinine sample (i.e., $7, $12, $17, and $22).
  3. A reset contingency will be used. That is the reward amount will be returned back to original $7 if there is a missing or positive saliva cotinine sample
Period: Overall Study
Arm/Group | Active Control | Media Literacy | Financial Incentive | Combined
Started | 9 | 11 | 10 | 10
Completed | 6 | 5 | 5 | 5
Not Completed | 3 | 6 | 5 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Control | Media Literacy | Financial Incentive | Combined | Total
Number analyzed (Participants) | 9 | 11 | 10 | 10 | 40
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 23 [22 to 28] | 25 [21 to 26] | 24 [23 to 25] | 22.5 [21 to 26] | 23.5 [22 to 26]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 7 | 9 | 7 | 7 | 30
  Male | 1 | 1 | 1 | 2 | 5
  Non-binary | 1 | 1 | 2 | 1 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 2 | 2 | 9
  Not Hispanic or Latino | 6 | 9 | 8 | 8 | 31
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 6 | 9 | 8 | 8 | 31
  Black | 0 | 2 | 2 | 2 | 6
  Other (e.g/., Asian or American Indian/Alaskan Native) | 0 | 0 | 0 | 0 | 0
  Unknown | 3 | 0 | 0 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 9 | 11 | 10 | 10 | 40

OUTCOME MEASURES:

1. Primary Outcome: Engagement_remote checkin_3
Description: Engagement will be assessed by proportions of participants who submitted the remote saliva cotinine sample at remote checkin 3.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Active Control | Media Literacy | Financial Incentive | Combined
Number analyzed (Participants) | 9 | 11 | 10 | 10
Participants
  Submitted | 6 | 5 | 6 | 5
  Missing | 3 | 6 | 4 | 5
Statistical Analysis 1: Comparison: Active Control vs Media Literacy vs Financial Incentive vs Combined; Test type: Superiority; p = 0.820, Fisher Exact

2. Primary Outcome: Retention
Description: The number of participants who completed the end-of-study assessment (Week 12).
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Active Control | Media Literacy | Financial Incentive | Combined
Number analyzed (Participants) | 9 | 11 | 10 | 10
Participants
  Completed | 6 | 5 | 5 | 5
  Missing | 3 | 6 | 5 | 5

3. Secondary Outcome: Biochemically Verified Vaping Abstinence
Description: Biochemically verified vaping abstinence (negative results- < 30 ng/mL) will be measured by saliva cotinine samples at end of study (Week 12).
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Active Control | Media Literacy | Financial Incentive | Combined
Number analyzed (Participants) | 9 | 11 | 10 | 10
Participants
  Postive | 2 | 0 | 0 | 2
  Negative | 4 | 5 | 5 | 3
  Missing | 3 | 6 | 5 | 5

4. Secondary Outcome: Self-reported Vaping Abstinence
Description: Self-reported vaping abstinence will be assessed by the question "In the past 30 days, did you vape at all, even a puff of someone else?" at the end-of-study visit.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Active Control | Media Literacy | Financial Incentive | Combined
Number analyzed (Participants) | 9 | 11 | 10 | 10
Participants
  Positive | 2 | 3 | 1 | 2
  Negative | 4 | 2 | 4 | 3
  Missing | 3 | 6 | 5 | 5

ADVERSE EVENTS:
Description: Given that our study included only behavioral interventions (text message support, media literacy education, and financial incentives), we did not collect adverse events, as the risk associated with the interventions was minimal.
Arm/Group | Active Control | Media Literacy | Financial Incentive | Combined
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-05-08): https://cdn.clinicaltrials.gov/large-docs/08/NCT05586308/Prot_SAP_000.pdf